CLINICAL TRIAL: NCT05514392
Title: Comparison of Electromyographic Threshold and Dynamic Balance After Single Leg Cycling Ergometer and Double Leg Cycling Ergometer Training in Healthy Adults
Brief Title: The Effect of Bicycle Ergometer Training on Balance and Emg Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: emgandbalance_cyclingergometer
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Exercise, Aerobic
Keywords: electromyography; balance; muscle fatigue; single leg cycling training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Receiving Single Leg Cycling Ergometer Training: First of all, an initial warm-up will be done with 40 watts of exercise intensity for 3 minutes. Exercise will be started with 80 watts of exercise intensity and will be increased by 40 watts every 3 minutes. Cycling cadence will be determined as a pedaling speed of 80 revolutions per minute and patients will be asked to keep their dominant leg on the pedal and keep their non-dominant leg on the ground. The exercise protocol will consist of 2 sets as 15 minutes of exercise + 1 minute of break + 15 minutes of exercise. During the exercise, the heart rate and oxygen saturation of the participants will be monitored by finger pulse oximetry. EMG measurements were taken at the beginning and end of the ergometer training.
  Interventions: Device: HP Cosmos Torqoalizer
- Receiving Double Leg Cycling Ergometer Training: First, a 3-minute initial warm-up will be done with an exercise intensity of 40 watts. The workout will begin with an exercise intensity of 80 watts and increase by 40 watts every 3 minutes. Cycling cadence will be determined as a pedaling rate of 80 revolutions per minute and patients will be asked to pedal with both legs. The exercise protocol will consist of 2 sets of 15 minutes of exercise + 1 minute of break + 15 minutes of exercise. During the exercise, the heart rate and oxygen saturation of the participants will be monitored by finger pulse oximetry. EMG measurements were taken at the beginning and end of the ergometer training.
  Interventions: Device: HP Cosmos Torqoalizer

INTERVENTIONS:
Device: HP Cosmos Torqoalizer — Participants will sign a consent form approved by the ethics committee. Height, weight, thigh length, leg length, foot length and kinematic foot length will be recorded before data collection. Ergometer positions will be adjusted according to participant preference. Participants will be invited to the Health Sciences University Physiotherapy and Rehabilitation Hall once. Before starting the exercise of the participants, muscle activity, balance assessment, leg fatigue will be evaluated. Participants will be made an exercise protocol. At the end of the exercise, necessary evaluations will be made again, and then the person will rest for 1 hour. After 1 hour, the exercise groups will change; Persons receiving single foot bicycle ergometer training will receive double foot bicycle ergometer training, and the group receiving double foot bicycle ergometer training will receive single foot bicycle ergometer training. Necessary evaluations will be repeated at the end of the training.

SUMMARY:
The study will contribute to answering the question of 'in which exercise types of single-leg and double-leg exercise protocols will affect whether fatigue occurs early or not, and muscle activations will occur. In response to this question, clinicians will prefer to focus on which type of exercise produces more muscle activation and late fatigue. Few studies have been done on single and double leg bicycle ergometers in the literature. From these studies; While examining the lactate and EMG threshold values after cycling ergometer training, another study compared the effectiveness of single and double leg cycling ergometers. In the literature, EMG and dynamic balance were not used in the comparison after single and double leg bicycle ergometer training. In this study, the effectiveness of single and double legged bicycle ergometers will be compared by looking at EMG and dynamic balance changes.

DETAILED DESCRIPTION:
In humans, one side of the body is often preferred over the other to perform voluntary motor actions. There is evidence that in bipedal cycling training, where both legs are simultaneously involved in the motor task, the dominant leg contributes more to the power produced than the non-dominant leg. The magnitude of asymmetries between both legs can vary (eg 1-40%) and depend on the variable of interest (eg power, torque, etc.), pedaling phase, intensity and cadence. Bicycle ergometer leg exercise has been applied in the literature as an assessment tool for motor function, aerobic training method and also for individuals. Cycling performance depends on the optimization of physiological, psychological and biomechanical parameters. There are already many studies on physiological or psychological performance parameters. The pedaling paradigm has many advantages. It minimizes postural control, is characterized by a restricted kinematic trajectory, requires less effort for training control, and shares a similar muscle activation pattern with walking. EMG is an indirect measure of muscle activity as it detects the electrical activity produced by the passage of a nerve impulse that causes an action potential in the muscle cell membrane. This potential consists of three phases: membrane depolarization, repolarization, and hyperpolarization period, which produces an electric field picked up by the EMG electrodes. Decomposition techniques have been applied to EMG signals to identify motor patterns of joint activation between muscle groups, called motor modules or muscle synergies. Each synergy is represented by a spatial component that reflects the composition of muscle co-activation and a temporal component that elicits modulus uptake throughout the execution of the movement. Successfully applied to different motor behaviors, this analysis supports the hypothesis of a low-dimensional modular organization at the central nervous system level. Muscle electrical activity is measured using electromyography (EMG). The amplitude of the EMG signal has a monotonic relationship with the number of activated muscle fibers and is therefore a good indicator of contraction intensity. In dynamic studies, the signals reaching the motor unit, which can be detected at the location of the electrode, overlap electrically and are observed as a bipolar signal with symmetrical negative and positive amplitude distribution. The signal obtained without filtering is called the "Raw signal", which consists of periods of contraction and relaxation. During the rest period, the baseline EMG is observed, which depends on many factors (quality of the amplifier, environmental noise, and the quality of the given sensing condition) and should not exceed line 3 if these factors are within appropriate limits. 5 microvolts (mV). During normal bipedal bicycle pedaling, when the leg extensor muscles are active during the first half of the 360̊ crank cycle, crank torque is mainly produced in the down phase of each leg while pedaling. For training and rehabilitation purposes, they sometimes engage in 1-leg pedaling with crank torque produced by only one leg, emphasizing the need for ipsilateral flexor activity in the upward movement of the foot to produce crank torque while pedaling and produce a smooth pedaling motion throughout. the entire crank cycle. Therefore, single-leg pedaling requires cyclists to change how they control. multiple extensor and flexor leg muscles during the crank cycle. Therefore, the 1-leg bike has been proposed as a training tool to improve pedaling performance and is used in clinical settings for rehabilitation. EMG studies with bicycle ergometer are insufficient in the literature. During this activity, there is no study in the literature comparing single-leg and double-leg exercises during single-leg cycling exercise, which is frequently used to prevent premature fatigue in leg muscles in chronic obstructive pulmonary patients. Although ergometer exercise is frequently used in rehabilitation treatment, it increases maximum oxygen uptake and muscle strength, decreases systolic and diastolic blood pressures, decreases body weight and body fat, improves cognitive function, balance function and muscle activity in the literature is limited. This study will contribute to answering this question that the exercise types of single-leg and double-leg exercise protocols will affect whether muscle activations occur early or not. In response to this question, clinicians will prefer to focus on which type of exercise produces more muscle activation and late fatigue. There have been a few studies in the literature on single and double leg bicycle ergometers. From these studies; Looking at the lactate and EMG threshold values after cycling ergometer training, another study compared the effectiveness of a single ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Absence of comorbid disease of orthopedic, neurological, cardiopulmonary system
* Participants who have not participated in another clinical trial in the last 1 month
* Participants with a Body Mass Index (BMI) below 30 kg/m2

Exclusion Criteria:

* Participants who had hip, pelvis, knee, ankle surgery in the last year
* Participants with leg length inequality
* Those with known balance disorders in the last three months due to vestibular disorders, pregnancy, concussion participants
* Participants taking any medication that may affect alertness or balance.
* During the study protocol, the participants did not comply with the requested requests.
* Presence of peripheral nerve dysfunctions and neurological disorders
* Presence of a previous injury to the feet or legs
* Prior surgery on the lower extremities
* Systemic discomfort
* Pain and other medical conditions that may affect postural control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Superficial Electromyographic (EMG) Measurement | Change from baseline emg values in 30 minutes
  In the dominant lower extremity to evaluate muscle activity, rectus femoris, surface EMG signals will be recorded with the Trigno Avanti Wireless Surface EMG System. While the participant is standing in hip neutral and knee extension, the adhesive EMG electrode will be placed on the reference motor point. Superficial EMG values will be recorded throughout the exercise. During the research, EMG will be recorded from the stimulated muscles by applying two electrodes to the skin for each muscle. The amplitude, duration and shape of the evoked muscle action potentials obtained will be reflected as a result. The amplitudes of the EMG signals will be evaluated. The method to be used when evaluating EMG signal amplitudes will be the raw EMG calculation. While evaluating the data, the computer package programs will benefit.
Static-Dynamic Balance Evaluation with Isokinetic Balance Device | Change from baseline static and dynamic balance values in 30 minutes
  Static and dynamic balance performances will be evaluated using the isokinetic balance measurement system. In this system, there is a sensor in the center of the platform that detects every angular movement and sends the information directly to the computer. For the static balance test, it will be ensured that they stand on both feet and on the right/left foot with eyes open (EO) and eyes closed (EC), respectively. The arms are positioned next to the body. Between each test measurement lasting 20 seconds, approximately 40 seconds of rest will be given. For the dynamic balance test, the difficulty level of the test will be set to "20". In the test, they will be asked to circle clockwise 5 times in 60 seconds without bending their knees within the limited area on the computer screen. The Patient Record database module enables the creation of clinical cards for each case. It facilitates the comparison of each case's own tests.
Static Balance Evaluation with One Leg Standing Balance Test | Change from baseline static balance values in 30 minutes
  This test will be used to evaluate balance status in our study. During the application, the person raises one foot while standing. From this moment on, the time is kept with the help of a stopwatch. As soon as the person's foot touches the ground again, the time is stopped.If the person can stand on one leg for 30 seconds, the test is over. If the time is between 10 seconds and 5 seconds, there is an imbalance. Even if it is less than 5 seconds, there is a risk of falling.

SECONDARY OUTCOMES:
Fatigue Impact Scale | Change from baseline fatigue scale values in 30 minutes
  It is used to measure the physical, cognitive and social effects of fatigue. It consists of a total of 40 questions, of which 10 are cognitive, 10 are physical and 20 are social scales. Each question scores between 1 and 4. The maximum total score is 160. Effect of fatigue not at all (0-32) / a little (33-64) / moderate (65-96) / significant (97- 128) / very important (129-160) problem. In our study, it will be used to evaluate the physical, cognitive and social effects of fatigue resulting from single-leg and double-leg cycling ergometer exercise.
Evaluation of Leg Fatigue with the Modified Borg Scale (MBS) | Change from baseline leg fatigue scale values in 30 minutes
  This scale was developed by Borg in 1970 to measure the effort expended during physical exercise. It is a scale that is frequently used to evaluate the severity of dyspnea on exertion and the severity of dyspnea at rest. It consists of ten items describing the severity of dyspnea according to their degrees. Defining the severity of dyspnea on the scale makes it easier for patients to apply. In the studies carried out; It is stated that MBS is a reliable scale for determining the severity of dyspnea at rest and exertion, and is associated with respiratory rate and pulmonary function tests. In addition, it is emphasized that MBS is superior to other scales in terms of long-term reproducibility and can be used to predict ventilatory reserves of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ARSLANCA, Principal Investigator — Saglik Bilimleri Universitesi; Beyza DURAK, Principal Investigator — Saglik Bilimleri Universitesi; Serra Nisa KIŞ, Principal Investigator — Saglik Bilimleri Universitesi; Sude Asya ALŞAN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park S, Caldwell GE. Muscular activity patterns in 1-legged vs. 2-legged pedaling. J Sport Health Sci. 2021 Jan;10(1):99-106. doi: 10.1016/j.jshs.2020.01.003. Epub 2020 Jan 20. PMID 33518019
- [Background] Raez MB, Hussain MS, Mohd-Yasin F. Techniques of EMG signal analysis: detection, processing, classification and applications. Biol Proced Online. 2006;8:11-35. doi: 10.1251/bpo115. Epub 2006 Mar 23. PMID 16799694
- [Background] Ambrosini E, De Marchis C, Pedrocchi A, Ferrigno G, Monticone M, Schmid M, D'Alessio T, Conforto S, Ferrante S. Neuro-Mechanics of Recumbent Leg Cycling in Post-Acute Stroke Patients. Ann Biomed Eng. 2016 Nov;44(11):3238-3251. doi: 10.1007/s10439-016-1660-0. Epub 2016 Jun 1. PMID 27251336